CLINICAL TRIAL: NCT02232048
Title: The Influence of Corticosteroid Treatment on Heart Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0061-14-HYMC
Record Dates: First submitted 2014-08-20; First posted 2014-09-04 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Corticosteroid Treatment: Patients in the internal medicine department who are being treated with corticosteroids will undergo Transthoracic Echocardiogram to determine change in heart function.
  Interventions: Other: Transthoracic Echocardiogram

INTERVENTIONS:
Other: Transthoracic Echocardiogram
  Other Names: Transthoracic Echocardiogram using a VIVID 6 device

SUMMARY:
Patients hospitalized in internal medicine departments are given corticosteroid treatment according clinical indications. Patients receive treatment at different dosage levels and in different preparations according to clinical indications. This study will investigate how corticosteroids effect the heart and specifically, longitudinal strain.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients able to undergo Transthoracic Echocardiogram
* Patients beginning treatment with corticosteroids

Exclusion Criteria:

* Pregnant
* Patients recently or chronically treated with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with corticosteroids for various clinical indications who have been hospitalized in the internal medicine department of the Hillel Yaffe Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Function | Two years
  Heart contraction and specifically its longitudinal strain will be examined using Transthoracic Echocardiogram (TTE) before, during and after corticosteroid treatment. TTE reveals changes in contraction in the right and left ventricle and septum.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel